CLINICAL TRIAL: NCT05036837
Title: OZOPROMAF: Validation Study of the Use of Ozonotherapy in Mronj Management- Protocol of Ozone by Infiltrations in Patients With Osteonecrosis of the Jaws Drug Related
Brief Title: Infiltration of Medical Ozone for the Treatment of Medication-Related Osteonecrosis of the Jaws (MRONJ)
Acronym: OZOPROMAF
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: DUE TO PANDEMIC CONDITIONS
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Olga Di Fede, Associate professor, University of Palermo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZOPROMAF_SEQ1
Record Dates: First submitted 2021-06-16; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: MEDICATION RELATED OSTEONECROSIS OF THE JAW
Keywords: MRONJ; Osteonecrosis; Jaw; Antiresorptive; Antiangiogenic drugs; Adverse event
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OZOPROMAF_SEQ1 (Experimental): OZOPROMAF consists of: local superficial anesthesia by application of EMLA® cream, intra-tissue injection of a 15 ml OxigenOzone (O2O3) mixture by 26Gx 1⁄2 - 0.45x13mm needle into mucosal margin surrounding bone exposure or around situs evidenced by CT scans.
  Pain intensity and/or other symptoms are assessed at each visit and the day after by a questionnaire (numerical rating scale).
  OZOPROMAF is applied on 7-15 days, depending on patient compliance, until the resolution (i.e. formation of sequestrum and clinical healing -T1).
  Follow-up visits are scheduled to confirm healing at 1 (T2), 3, 6 (T3), 12 (T4), 18- 24 months (T5). Radiographic evaluations of bone healing are scheduled at T3/ T4/T5.
  Positive outcomes
  at T1/T2 clinical healing (no signs of acute phlogosis and no symptoms compatible with MRONJ);
  at T3/ T4/T5 clinical healing and no radiological signs of MRONJ.
  Interventions: Drug: OZOPROMAF_SEQ1

INTERVENTIONS:
Drug: OZOPROMAF_SEQ1 — OZOPROMAF protocol consists of: local superficial anesthesia by EMLA® cream, intra-tissue injection of a 15 ml OxigenOzone (mixture by 26Gx 1⁄2 - 0.45x13mm needle into the mucosal margin surrounding the bone exposure or around the situs already evidenced by CT scan. It is applied on 7-15 days, depending on the patient compliance, until the formation of sequestrum and clinical healing (T1).
  Pain intensity is assessed by means of a questionnaire for pain and/or other symptoms evaluation before and after the protocol, based on numerical rating scale (NRS).
  After resolution (T1), follow-up visits are scheduled to confirm the healing of MRONJ at 1 (T2), 3, 6 (T3), 12 (T4), 18- 24 months (T5).
  Radiographic evaluations of bone healing are scheduled at T3 and T4.
  Positive outcomes for the OZOPROMAF protocol are evaluated at T1 as no clinical signs of acute phlogosis and no symptoms compatible with MRONJ; at T5 as clinical healing and no radiological signs of MRONJ.

SUMMARY:
Medication-related osteonecrosis of the jaw (MRONJ) is a serious adverse reaction of antiresorptive and antiangiogenic agents; it is also a potentially painful and debilitating condition. Today, no specific studies have prospectively evaluated the efficacy of its treatment and no robust standard of care has been established.

Among non-invasive procedures to treat MRONJ, the use of medical ozone (O3) arises for its properties and has been deployed and evaluated. O3 has generally proven to play a role in the treatment of chronic, nonhealing, or ischemic wounds, due to its antimicrobial and anti-oxidant properties and to bio-stimulation; it has been extensively used for different medical approaches and purposes. In oral cavity, local applications are carried out by ozonized water (i.e. spray or compress) or gel.

The aim of this open trial is to assess the efficacy and the safety of O3 by a new method of application, i.e. infiltrations of oral mucosa, in patients with a diagnosis of MRONJ, which are non-eligible for the standard of care, regardless staging.

All cases included in our study are MRONJ and staged according to the classification of the Italian Societies of Oral Medicine and Maxillofacial Surgery (the SICMF/SIPMO staging system); in addition, they arereported to AIFA, the Italian Medicines Agency, for registration of the adverse event drug related.Patients included in our study are selected due to their non-eligibility to the standard treatment (conservative/medical for long term or surgical alone) for unstable systemic conditions or unaccepted consent due to extensive proposed approach due to the advanced disease.

During the first examination (T0), medical, pharmacological, and dental history of patients are recorded. Data collected are: (1) age; (2) gender; (3) indications for use, type, cumulative dose and duration of MRONJ-related drugs; (4); history of chemotherapy; (5) other medications; (6) other diseases; (7) smoking.

For every patient, Cone Beam CT dental scan or maxillofacial CT scan has performed for staging at T0 and 12 (T4) months after; orthopantomograph has performed during protocol (T3). The main CT features evaluated and associated to MRONJ presence and healing are as follows: a) bone sclerosis, b) depth of lesion; c) formation of sequestrum.

When more than one MRONJ lesion are present, the protocol is applied one by one.

DETAILED DESCRIPTION:
OZOPROMAF protocol consists of: local superficial anesthesia by application of EMLA® cream, intra-tissue injection of a 15 ml OxigenOzone (O2O3) mixture by 26Gx 1⁄2 - 0.45x13mm needle into the mucosal margin surrounding the bone exposure or around the situs already evidenced by CT scan.

Moreover, pain intensity is assessed at each visit by means of a questionnaire for pain and/or other symptoms evaluation before and after the protocol, based on numerical rating scale (NRS).

OZOPROMAF is applied on 7-15 days, depending on the patient compliance, until the resolution, identified as formation of sequestrum and clinical healing (T1).

The day after the procedure, every patient iss supported by phone evaluating pain and/or adverse events with a questionnaire In case of unavailability of the patient for the weekly treatment, it is mandatory the phone call for the questionnaire, in order to evaluate symptoms by simple questions and NAS scale.

After resolution (T1), follow-up visits are scheduled to confirm the healing of MRONJ at 1 (T2), 3, 6 (T3), 12 (T4), 18- 24 months (T5). Radiographic evaluations of bone healing are scheduled at T3 and T4.

Positive outcomes for the OZOPROMAF protocol are evaluated at T1 as no clinical signs of acute phlogosis and no symptoms compatible with MRONJ; at T5 as clinical healing and no radiological signs of MRONJ.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of MRONJ
* Patients with MRONJ non-eligibilible to the standard treatment (medical or surgical alone) for unstable systemic conditions or for unaccepted consent due.

Exclusion Criteria:

* Head and neck radiotherapy
* Long term sistemic antimicrobial therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
MUCOSAL HEALING | 3 months
  no clinical signs and no symptoms compatible with MRONJ outcome measure:
  * formation of sequestrum by visualization of bone sequestrum
  * no infectius signs by visual inspection
  * no pain by NAS
MUCOSAL HEALING (1-T2) | 3 months (T2)
  no clinical signs Outcome measure: no clinical signs compatible with MRONJ by visual inspection
MUCOSAL HEALING (2-T2) | 3 months (T2)
  no symptoms Outcome measure: pain evaluation by NAS
BONE HEALING (T2) | 3 months (T2)
  Outcome measure: no radiological signs compatible with MRONJ by OPT (orthopantomograph)
MUCOSAL HEALING (1-T3) | 6 months (T3)
  no clinical signs Outcome measure: no clinical signs compatible with MRONJ by visual inspection
MUCOSAL HEALING (2-T3) | 6 months (T3)
  no symptoms Outcome measure:pain evaluation by NAS
BONE HEALING (T3) | 6 months (T3)
  Outcome measure: no radiological signs compatible with MRONJ by CT (computed tomography)
MUCOSAL HEALING (1-T4) | 12 months (T4)
  no clinical signs Outcome measure: no clinical signs compatible with MRONJ by visual inspection
MUCOSAL HEALING (2-T4) | 12 months (T4)
  no symptoms Outcome measure:pain evaluation by NAS
BONE HEALING (T4) | 12 months (T4)
  Outcome measure:
  no radiological signs compatible with MRONJ by CT (computed tomography)
MUCOSAL HEALING (1-T5) | 18-24 months (T5)
  no clinical signs Outcome measure: no clinical signs compatible with MRONJ by visual inspection
MUCOSAL HEALING (2-T5) | 18-24 months (T5)
  no symptoms Outcome measure: pain evaluation by NAS
BONE HEALING (T5) | 18-24 months (T5)
  Outcome measure:
  no radiological signs compatible with MRONJ by CT (computed tomography)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Di Fede, Professor, Principal Investigator — University of Palermo - Italy
Locations (1):
- Azienda Ospedaliera Universitaria Policlinico "P. Giaccone" Palermo - University of Palermo, Palermo, Italy - Sicily, Italy

IPD SHARING:
Plan to Share IPD: Yes
Patients included in our study are selected due to their non-eligibility to the standard treatment (conservative/medical for long term or surgical alone) for unstable systemic conditions or unaccepted consent due to extensive proposed approach due to the advanced disease.
Supporting Information: Study Protocol

REFERENCES:
- See also: Related Info — https://giuseppinacampisi.it/promaf/